CLINICAL TRIAL: NCT00230425
Title: The Measurement of Mood Variability and Sustained Attention in Women With Alcohol Dependence.
Status: Completed | Type: Observational
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatoon Health Region (Other)
Other Study IDs: BSC 02-760
Record Dates: First submitted 2005-09-27; First posted 2005-09-30 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2005-09

CONDITIONS: Alcohol Abuse; Anxiety Disorders; Mood Disorders
Keywords: Alcohol Abuse; Anxiety Disorders; Mood Disorders
MeSH Terms: conditions — Alcoholism; Anxiety Disorders; Mood Disorders

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this study is to measure daily mood changes and to find out whether these mood changes are related to the ability to maintain attention on a task. Problems with mood are more common among women however, the association between symptoms of alcohol abuse and mood syndromes is inconsistent.

First we hypothesize that women with lifetime diagnoses of alcohol abuse will not demonstrate higher symptoms of anxiety, depression, neuroticism and mood variability than control groups. Second, that the severity of these symptoms will not correlate with performance on measures of sustained attention.

DETAILED DESCRIPTION:
Epidemiological and clinical studies show an association between symptoms of anxiety and depression (mood) and alcohol abuse. However, the association between alcohol abuse and mood syndromes is inconsistent. One problem is that mood syndromes tend to be poorly defined. Also, researchers typically have relied on retrospective recall by patients to evaluate mood symptoms.

Some of this evidence is that:

1. Most mood symptoms improve with withdrawal in inpatient alcoholism programs without specific treatment of the mood disorder.
2. Family genetic studies have not shown cosegregation.
3. Psychiatric treatment of mood syndromes does not decrease alcohol use.
4. The self-treatment view has not been supported by controlled drinking studies.

To overcome this difficulty, we have recently developed a procedure to measure mood variability while it is occurring. We ask participants to rate their moods twice a day on a 10 cm straight line anchored by the terms "not at all" and "very much so" (a visual analogue scale) (VAS). There are 3 separate lines for "anxiety/tension", "sadness/low mood" and "high mood". We then compute a quantitative measure of variability the "mean squared successive difference statistic" (MSSD). Our earlier work found that this method identified greater mood variability in individuals with anxiety disorders as compared to individuals without anxiety disorders.

Our null hypotheses are:

1. That women with lifetime diagnoses of alcohol abuse will not demonstrate higher symptoms of anxiety, depression, neuroticism and mood variability than control groups and;

1a. That the severity of these symptoms will not correlate with performance on measures of sustained attention.

The MINI diagnostic interview will be used to derive DSM-IV diagnoses. This is a brief semi-structured diagnostic interview that we have used previously. We have not used an extensive interview schedule such as the SCID because we are not recruiting specific diagnostic groups.

Participants will be asked to complete 4 scales as validators of the diary visual analogue scales. These are:

1. The Beck Depression Inventory (BDI-II). This is the most widely used self- completed depression questionnaire. It has 21 items, each has 4 choices.
2. The Spielberger Trait-State Self-Evaluation Questionnaire (STAI-T). This is a 20 item- questionnaire, with answers on a 4-point scale. It is the most widely used trait anxiety inventory.
3. The Mood Disorders Questionnaire. This is a recently developed but well researched questionnaire to measure high mood. Sixteen questions are in a yes/no format.
4. 12 items from the Neuroticism Scale of the Eysenck Personality Inventory as modified by Kendler. These items are answered yes/no.

Participants will be females, aged 18-50 years with diagnoses of alcohol abuse. Exclusion criteria will be chronic medical, psychiatric or brain conditions that might affect mood variability or test performance. Comorbid drug abuse will not be reason for exclusion.

Only females are included in this study because

1. The association between mood symptoms and substance abuse appears to be clearer in women (In men, other characteristics such as impulsivity and antisocial traits are more prominent).
2. We already have data on mood variability in predominantly female normal control subjects from studies in the Department of Psychiatry at Royal University Hospital.

Participants will be tested in their 3rd and 4th weeks of the program, i.e. they will have been free of alcohol and illicit drug consumption for 3 weeks. Use of other medication will be noted but will not be an exclusion.

ELIGIBILITY:
Inclusion Criteria:

* Females ages 18 to 50.
* Diagnosed with alcohol abuse issues.

Exclusion Criteria:

* Males (any age).
* Chronic medical (organic) or psychiatric conditions that might affect mood variability or test performance.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 2003-02; Study Completion 2004-06

CONTACTS AND LOCATIONS:
Overall Officials: Rudy Bowen, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Calder Centre, Saskatoon, Saskatchewan, Canada